CLINICAL TRIAL: NCT05205876
Title: A Safety and Feasibility Study of the Eddii Mobile Application for Glucose Monitoring in Pediatric Patients With Type I Diabetes
Brief Title: Safety and Feasibility Study of the Eddii Mobile Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eddii, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LeafStudy
Record Dates: First submitted 2021-12-10; First posted 2022-01-25 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Type-1 Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Dexcom app) (No Intervention): This group will use the Dexcom application for management of their blood glucose for the duration of the study (8 weeks).
- Intervention (Eddii app) (Experimental): This group will use the Dexcom application for the initial 2 weeks of the study, and switch to using the Eddii application on Day 14 of the study for the remaining 6 weeks of the study.
  Interventions: Behavioral: Eddii mobile application

INTERVENTIONS:
Behavioral: Eddii mobile application — Participants will use the Eddii mobile application in the intervention arm.
  Arms: Intervention (Eddii app)

SUMMARY:
The study is designed to measure the safety and feasibility of the Eddii mobile app for children living with Type-1 diabetes and using a CGM (Continuous Glucose monitor).

DETAILED DESCRIPTION:
Wearable continuous glucose monitoring (CGM) sensors have revolutionized diabetes management over the past decade. By providing blood glucose (BG) concentration measurements continuously over consecutive days, CGMs are an increasingly adopted technology. While CGM devices have been shown to improve the safety and effectiveness of diabetes therapy to reduce hypoglycemia incidents and durability and to decrease glycemic variability CGM software and tools available for users to feel motivated and engaged are limited. Users of CGM often use an app that provides an interface for them to track their BG. In most cases, this app is offered by their CGM device provider.

These interfaces are considerably basic and scientific in nature, often developed by scientists and engineers for the everyday user. These apps are particularly dull and tiresome for children and adolescents living with diabetes. Current real-time CGM interfaces present real-time BG reading, in addition to the BG trend and a historical chart, together with minimal options for the user to enter lifestyle data such as medications, meals, and exercise. Examples of such default interfaces are ones offered by Dexcom, Medtronic Guardian and Freestyle Libre. While some of these apps provide patterns and health summaries to the user, these are provided in a separate app to the one streaming real-time BG. With the emergence of rtAPI (real-time Application Programming Interface) integrations with CGMs, there is ample opportunity to improve the dynamism, sophistication, and offerings within these CGM Apps , creating a platform that delights the user rather than one that makes diabetes management seem like a daily chore. Furthermore, it is hypothesized that creating additional engagement in the form of games and real-life rewards will improve glycemic control.

ELIGIBILITY:
Inclusion Criteria (Pediatric Volunteers)

Subject must meet all of the following to be enrolled.

* Volunteer, or their Authorized Representative, is willing and able to provide written informed consent, including authorization to release health information
* Volunteer is > 5 years and < 12 years of age (inclusive) at time of consent
* Volunteer has been diagnosed with Type 1 diabetes
* Volunteer has been utilizing the Dexcom continuous glucose monitor for a minimum of 6 months prior to enrollment in the study
* Volunteer must use the Dexcom mobile application
* Volunteer has a parent or legal guardian willing to participate in the study
* Volunteer must have access to and use an iOS smart phone, iPhone 10 model or above

Parent / Guardian Volunteers:

Subject must meet all of the following to be enrolled.

* Volunteer is willing and able to provide written informed consent, including authorization to release health information
* Volunteer has a child that meets study inclusion criteria and is willing to participate in the study
* Volunteer lives with a child that meets study inclusion criteria and is willing to participate in the study
* Volunteer is willing to be responsible for management of the Eddii mobile application use
* Volunteer must have and use an iOS smart phone device

Exclusion Criteria:

- EXCLUSION CRITERIA (Pediatric Volunteers)

Subject will be excluded if any of the below are present.

* Volunteer is unwilling or unable to provide written informed consent and/or does not have an authorized representative who can provide consent on their behalf
* Volunteer does not have access to an iOS smartphone device
* Volunteer does not have access to the internet
* Volunteer is enrolled in another research study at the time of enrollment

EXCLUSION CRITERIA (Parents / Guardians) Subject will be excluded if any of the below are present.

* Volunteer is unwilling or unable to provide written informed consent and/or does not have an authorized representative who can provide consent on their behalf
* Volunteer does not have access to an iOS smartphone device
* Volunteer does not have access to the internet
* Volunteer is enrolled in another research study at the time of enrollment

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Safety of the Eddii App as assessed by accuracy and reliability of blood glucose measurements | Eight Weeks
  Safety (Intervention Arm only) as assessed by:
  ○ Functionality and reliability of Eddii application by measuring reported faults
Feasibility of the Eddii App as measured by frequency of use | Four Weeks
  Feasibility (Intervention Arm only) as measured by:
  * App analytics to determine total number and frequency of logins from enrollment to Week 8
  * App analytics to determine application features are easily accessible, understandable and are used effectively

SECONDARY OUTCOMES:
Change in glycaemic control measured as Time-in-Range (TIR) (70-180mg/dl) | Eight Weeks
QOL (Quality of Life) metrics | Eight Weeks
  - QOL questionnaires conducted mid-study on weeks 2, 4, 6 and 8
User Engagement measured through app analytics | Eight Weeks
  App-Specific Measures for Entirety of Study (Intervention Arm only)
  ○ Engagement and retention of users

CONTACTS AND LOCATIONS:
Overall Officials: Farhaneh Ahmadi, PhD, Principal Investigator — Eddii, Inc.
Locations (1):
- Eddii, inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No